CLINICAL TRIAL: NCT07031388
Title: Effectiveness of HydrogenPeroxie, Hyaluronic Acid, Chlorhexidine Mouthwashes in Gingivitis Management: A Randomized, Triple-Blind, Controlled Clinical Trial
Brief Title: Mouthwashes for Gingivitis: Comparing a Hydrogen Peroxide-Hyaluronic Acid Mix, Hyaluronic Acid, and Chlorhexidine, A Triple-Blind Clinical Trial
Acronym: TRIPLE-G
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ramziyah Hayder Bakr (Other)
Responsible Party: Sponsor-Investigator, Ramziyah Hayder Bakr, Board Candidate in Dental Public Health, Kurdistan Higher Council of Medical Specialties
Organization: Kurdistan Higher Council of Medical Specialties (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RP-DPH-KHCMS-2025-001
Record Dates: First submitted 2025-05-28; First posted 2025-06-22 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Plaque Induced Gingival Disease
Keywords: Triple blind clinical trial; Gingivitis; Hydrogen peroxide; Hyaluronic acid; Chlorhexidine
MeSH Terms: conditions — Gingivitis | interventions — Hyaluronic Acid; Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of four parallel treatment groups, each receiving a different mouthwash intervention for gingivitis management.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1- Arm 1 Hydrogen peroxide + Hyaluronic acid (Experimental): Participants in this arm will receive a mouthwash formulation containing 1.8% hydrogen peroxide and 0.10% hyaluronic acid. The mouthwash is to be used twice daily for 3 weeks, following standardized oral hygiene instructions. This combination is intended to synergize the antimicrobial effects of hydrogen peroxide with the anti-inflammatory and healing properties of hyaluronic acid to manage gingivitis.
  Interventions: Combination Product: 1-Hydrogen peroxide and hyaluronic acid
- 2- Arm 2 Hyaluronic acid alone (Experimental): Participants in this arm will use a mouthwash containing 0.12% high molecular weight hyaluronic acid only. The mouthwash will be used twice daily for 3 weeks. Hyaluronic acid is known for its anti-inflammatory, tissue repair, and moisturizing effects, and this arm will assess its standalone effectiveness in improving gingival health in patients with gingivitis.
  Interventions: Combination Product: 2- Hyaluronic acid
- 3- Arm 3 chlorhexidine (CHX) (Experimental): Participants in this arm will receive a commercially available mouthwash containing 0.12% chlorhexidine gluconate. The solution will be used twice daily for 3 weeks, following standardized oral hygiene instructions. Chlorhexidine is a widely used antiseptic known for its broad-spectrum antimicrobial activity and effectiveness in reducing plaque and gingival inflammation.
  Interventions: Combination Product: Chlorhexidine
- 4- Arm 4 placebo (Placebo Comparator): Participants in this arm will receive a placebo mouthwash designed to closely mimic the active treatments in appearance, taste, and viscosity, ensuring effective blinding. The formulation comprises:
  * 2 ml glycerin
  * Vanilla flavoring agent
  * Brown food coloring
  * Distilled water to make up 1 liter
  This placebo was prepared at Awamedica, a certified Class A pharmaceutical manufacturer known for its state-of-the-art formulation laboratory and commitment to quality in pharmaceutical manufacturing. The solution is dispensed in 120 ml opaque brown bottles, each labeled solely with the participant's number to maintain blinding. Participants are instructed to use the mouthwash twice daily for 3 weeks, following standardized oral hygiene instructions. This arm serves as a negative control to assess the true efficacy of the active mouthwash formulations in managing gingivitis.
  Interventions: Combination Product: Placebo mouthwash

INTERVENTIONS:
Combination Product: 1-Hydrogen peroxide and hyaluronic acid — Hydrogen Peroxide (1.80%): Acts as an antiseptic agent, releasing oxygen that helps in reducing bacterial load and disrupting biofilms associated with gingivitis.
  * Hyaluronic Acid (0.10%): A naturally occurring polysaccharide known for its anti-inflammatory and tissue-regenerative properties, aiding in the healing of gingival tissues Clinical studies have demonstrated the efficacy of Perhyal in managing gingivitis. In a randomized controlled trial, Perhyal showed a significant reduction in gingival inflammation compared to placebo, with no reported adverse effects over 21 days.
  Arms: 1- Arm 1 Hydrogen peroxide + Hyaluronic acid
Combination Product: 2- Hyaluronic acid — This intervention involves the use of a mouthwash containing hyaluronic acid (0.12%) of high molecular weight, without any additional active agents. Hyaluronic acid is a naturally occurring substance known for its anti-inflammatory and wound-healing properties. It supports gingival tissue regeneration and hydration, which may contribute to reducing signs of gingivitis such as redness, swelling, and bleeding. Participants assigned to this arm will rinse with 10 mL of the solution twice daily for three weeks, following standardized oral hygiene instructions. This arm serves to evaluate the independent therapeutic effect of hyaluronic acid in managing gingival inflammation.
  Arms: 2- Arm 2 Hyaluronic acid alone
Combination Product: Chlorhexidine — This intervention uses a commercially available chlorhexidine gluconate 0.12% mouthwash, widely recognized for its strong antimicrobial properties. Chlorhexidine is considered a gold-standard agent for chemical plaque control and is effective in reducing bacterial load, gingival inflammation, and bleeding. Participants in this group will rinse with 10 mL of the solution twice daily for three weeks, in addition to maintaining regular oral hygiene practices.
  Arms: 3- Arm 3 chlorhexidine (CHX)
Combination Product: Placebo mouthwash — This placebo mouthwash was specially formulated to visually and sensorially resemble the active mouthwash products without containing any active therapeutic ingredients. It was prepared in the AwaMedica laboratory using 1 liter of distilled water, 98.5% distilled water, 2 mL of glycerin for mild viscosity, 5 mL of vanilla flavoring for taste masking, and 8 mL of brown food coloring to match the appearance of chlorhexidine. The solution was stored in 120 mL opaque brown bottles, each labeled only with the participant number to ensure blinding. Participants will use 10 mL of the placebo rinse twice daily for three weeks, following the same oral hygiene protocol as other groups.
  Arms: 4- Arm 4 placebo

SUMMARY:
This randomized, triple-blind clinical trial is designed to evaluate the efficacy of four different mouthwash formulations - hydrogen peroxide with hyaluronic acid, hyaluronic acid alone, chlorhexidine, and placebo - in four parallel arms. The study will take place at multiple centers, starting on June 1, 2025, and is expected to conclude by October 1, 2026. There is no external funding source for this study.

Eligible participants include systemically healthy individuals aged 18 to 35 years with a gingival and plaque index score of 1 or higher. Individuals with systemic or oral diseases will be excluded. Participants will be randomly assigned to one of four groups, each receiving a different mouthwash formulation for twice-daily use, following standardized oral hygiene instructions.

The potential benefit includes a reduced risk of gingivitis progression to periodontitis. There are no significant anticipated risks, though mild oral discomfort or taste alteration may occur.

DETAILED DESCRIPTION:
This randomized, triple-blind clinical trial aims to compare the effectiveness and safety of four different mouthwash formulations in managing gingivitis. The test group will use a mouthwash containing hydrogen peroxide (H2O2 1.80% )and hyaluronic acid (HA 0.10%). The three comparator groups will receive either chlorhexidine (CHX 0.12%), hyaluronic acid (HA 0.12%) (high molecular weight) alone, or a placebo mouthwash.

A total of four parallel arms will be used. Participants will be randomly assigned using a computer-generated randomization list. Blinding will apply to participants, clinical evaluators, and data analysts to maintain objectivity (triple-blind design).

Each participant will use the assigned mouthwash twice daily for three weeks, following standard oral hygiene instructions.

The primary outcomes will be changes in gingival inflammation, plaque accumulation, and bleeding on probing, assessed using the Gingival Index (GI), Plaque Index (PI), and Bleeding on Probing (BOP). Measurements will be taken at baseline, and after one, two, and three weeks of intervention.

The secondary outcomes will include reported side effects such as taste alteration, tooth discoloration, and overall comfort using the mouthwash.

The study is designed to determine which formulation offers the best balance of clinical effectiveness and patient acceptability in gingivitis management.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a gingival index score of 1 or greater.
* Subjects with a plaque index score of 1 or greater
* Systemically healthy individuals.
* Minimum of 20 natural teeth

Exclusion Criteria:

* Current use of any mouthwash.
* Smoking habit.
* Presence of active caries.
* Overhanged restorations and crowns.
* Presence of supra or subgingival calculus.
* Ongoing orthodontic treatment (including post-treatment retainer)
* Periodontal treatment within the past 6 months and a diagnosis of periodontitis.
* Use of antibiotics within the past 4 months or requirement for antibiotic prophylaxis.
* Systematic or topical non-steroidal anti-inflammatory drug treatment for the past 4 months
* Pregnancy or lactation.
* History of heart valve replacement.
* Known intolerance or allergy to mouth rinses.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Gingival Index (GI) from baseline to week 3 | Baseline, Week 1, Week 2, Week 3
  Mean Gingival Index score per participant, assessed on six sites per tooth. Score range: 0 (normal) to 3 (severe inflammation).
Change in Plaque Index (PI) from baseline to week 3 | Baseline, week 1, week 2, week 3
  Mean Plaque Index score per participant, assessed using the Silness and Löe method-score range: 0 (no plaque) to 3 (abundant plaque).
Change in Bleeding on Probing (BOP) from baseline to week 3 | baseline, week 1, week 2, week 3
  Percentage of sites showing bleeding on probing, recorded within 30 seconds after probing. Range: 0% to 100%.

SECONDARY OUTCOMES:
Change in Discomfort score after mouthwash use | After 3 weeks of mouthwash use
  Discomfort will be assessed using a Visual Analog Scale (0 = no discomfort, 10 = extreme discomfort). A higher score indicates worse discomfort.
Change in taste perception after mouthwash use | After 3 weeks of mouthwash use
  Presence or absence of taste change (yes/no)
  * Type of alteration (metallic, bitter, sweet, sour, salty, other)
  * Intensity (mild, moderate, severe)
  * Duration (less than 5 minutes, 5-15 minutes, 15-30 minutes, more than 30 minutes)
Change in tooth color shade assessed by VITA easy shade LITE | At baseline and after 3 weeks of mouthwash use
  Tooth color will be assessed at baseline and the end of the study using a VITA shade guide (VITA easy shade LITE). Shade values (e.g., A3, B1, 1L1.5, 2L1.5) will be recorded as observed. Changes will be presented as direct comparisons between baseline and final visit for each participant (e.g., "A3 to B1").
  No numerical scale or categorization will be applied. The results will be reported as the exact shade code changes observed using the VITA system.

CONTACTS AND LOCATIONS:
Locations (1):
- khanzad specialized health centre + Hwler dental center + Azadi dental center + Students of Hawler medical college, Erbil, Kurdistan, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing has not been confirmed at this stage. It depends on future institutional decisions and ethical approvals.